CLINICAL TRIAL: NCT03358472
Title: A Phase 3 Randomized, Open-Label Clinical Study to Evaluate the Efficacy and Safety of Pembrolizumab Plus Epacadostat, Pembrolizumab Monotherapy, and the EXTREME Regimen as First Line Treatment for Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (KEYNOTE-669/ECHO-304)
Brief Title: Pembrolizumab Plus Epacadostat, Pembrolizumab Monotherapy, and the EXTREME Regimen in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (KEYNOTE-669/ECHO-304)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEYNOTE-669/ECHO 304; 2017-001338-24 (EudraCT Number)
Record Dates: First submitted 2017-11-27; First posted 2017-11-30 (Actual); Results first posted 2019-09-10 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck squamous cell carcinoma; programmed cell death 1 (PD-1) inhibitor; indoleamine 2,3-dioxygenase 1 (IDO1) inhibitor
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; epacadostat; Cetuximab; Cisplatin; Carboplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab + Epacadostat (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: Epacadostat
- Pembrolizumab (Experimental)
  Interventions: Drug: Pembrolizumab
- EXTREME (Active Comparator): EXTREME regimen includes cetuximab + cisplatin or carboplatin + 5-fluorouracil.
  Interventions: Drug: Cetuximab; Drug: Cisplatin; Drug: Carboplatin; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab administered intravenously every 3 weeks.
  Other Names: MK-3475
  Arms: Pembrolizumab; Pembrolizumab + Epacadostat
Drug: Epacadostat — Epacadostat administered orally twice daily.
  Other Names: INCB024360
  Arms: Pembrolizumab + Epacadostat
Drug: Cetuximab — Cetuximab administered intravenously on Cycle 1 Day 1 followed by administration every week.
  Arms: EXTREME
Drug: Cisplatin — Cisplatin administered intravenously every 3 weeks for </= 6 cycles.
  Arms: EXTREME
Drug: Carboplatin — Carboplatin administered intravenously every 3 weeks for </= 6 cycles.
  Arms: EXTREME
Drug: 5-Fluorouracil — 5-Fluorouracil administered intravenously every 3 weeks for </= 6 cycles.
  Arms: EXTREME

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of pembrolizumab plus epacadostat, pembrolizumab monotherapy, and the EXTREME regimen (cetuximab + cisplatin or carboplatin + 5-fluorouracil) as first-line treatment for recurrent or metastatic head and neck squamous cell carcinoma (HNSCC).

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease based on RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function per protocol-defined criteria.
* Documentation of results from testing of human papilloma virus (HPV) status for oropharyngeal cancer.
* Baseline archival tumor specimen available or willing to undergo a prestudy treatment tumor core or excisional biopsy of a tumor lesion not previously irradiated, to obtain the specimen.

Exclusion Criteria:

* Carcinoma of the nasopharynx, salivary gland, unknown primary origin, or nonsquamous histologies as primary tumors.
* Disease progression within 6 months of completion of curatively intended systemic treatment for locoregionally advanced HNSCC.
* Use of protocol-defined prior/concomitant therapy.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Active autoimmune disease that has required systemic treatment in past 2 years.
* Known history of human immunodeficiency virus (HIV) infection. HIV testing is not required unless mandated by local health authority.
* Known history of or is positive for active hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (defined as HCV RNA [qualitative] is detected).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2025-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jones, MD, Study Director — Incyte Corporation
Locations (73):
- United States (14):
  - Pacific Cancer Medical Center, Anaheim, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Northwest Georgia Oncology Centers PC, Douglasville, Georgia
  - U of Kansas Cancer Center, Westwood, Kansas
  - Baptist Health, Louisville, Kentucky
  - St. Vincent Healthcare Cancer Ctr, Billings, Montana
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Oklahoma Cancer Specialists and Research, Tulsa, Oklahoma
  - Providence Portland Med Center, Portland, Oregon
  - Huntsman Cancer Institute Univ of Utah, Salt Lake City, Utah
  - Viginia Mason Med Ctr, Seattle, Washington
- Australia (3):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - Macquarie University Hospital, North Ryde, New South Wales
  - Royal Brisbane & Women s Hospital, Herston, Queensland
- Austria (2):
  - Landeskrankenhaus Salzburg, Salzburg
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
- Canada (4):
  - Juravinski Cancer Center Hamilton Health Sciences, Hamilton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-Universite Laval-Hotel Dieu de Quebec, Québec, Quebec
- Hungary (2):
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointezet, Szolnok
- Italy (2):
  - Istituto Europeo di Oncologia, Milan
  - IRRCS Instituto Clinico Humanitas, Rozzano
- Japan (14):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Miyagi Cancer Center, Natori-shi, Miyagi
  - Tohoku University Hospital, Sendai, Miyagi
  - Hyogo Cancer Center, Akashi
  - Kyushu University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Hokkaido University Hospital, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe
  - Saitama Cancer Center, Saitama
  - Kindai University Hospital, Sayama
  - Shizuoka Cancer Center Hospital and Research Institute, Shizuoka
  - The Cancer Institute Hospital of JFCR, Tokyo
- Poland (3):
  - Mazowiecki Szpital Onkologiczny, Wieliszew, Masovian Voivodeship
  - Przychodnia Lekarska Komed, Konin
  - Zachodniopomorskie Centrum Onkologii, Szczecin
- Portugal (4):
  - Inst. Portugues de Oncologia de Coimbra Frencisco Gentil EPE, Coimbra
  - Inst. Portugues de Oncologia de Lisboa Francisco Gentil EPE, Lisbon
  - Centro Hospitalar Lisboa Norte EPE - Hospital de Santa Maria, Lisbon
  - Inst. Portugues de Oncologia de Porto Francisco Gentil EPE, Porto
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (7):
  - Hospital Germans Trias i Pujol. ICO de Badalona, Badalona
  - Hospital General Universitari Vall d Hebron, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Infanta Cristina, Madrid
  - Hospital de Nuestra Senora de Valme, Seville
  - Hospital Clinico Lozano Blesa, Zaragoza
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation. Linkou, Taoyuan District
- Turkey (Türkiye) (7):
  - Adana Sehir Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Trakya Universitesi Tip Fakultesi, Edirne
  - Istanbul Universitesi Onkoloji Enstitusu, Istanbul
  - Medipol Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Inonu Universitesi Turgut Ozal Tip Merkezi, Malatya
- United Kingdom (5):
  - North Middlesex Hospital, London
  - University College London Hospitals (UCLH), London
  - The Royal Marsden Foundation Trust, London
  - The Royal Marsden Nhs Foundation Trust - Chelsea, London
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho BC, Brana I, Cirauqui B, Aksoy S, Couture F, Hong RL, Miller WH Jr, Chaves-Conde M, Teixeira M, Leopold L, Munteanu M, Ge JY, Swaby RF, Hughes BGM. Pembrolizumab plus epacadostat in patients with recurrent/metastatic head and neck squamous cell carcinoma (KEYNOTE-669/ECHO-304): a phase 3, randomized, open-label study. BMC Cancer. 2024 Jul 25;23(Suppl 1):1254. doi: 10.1186/s12885-023-11316-0. PMID 39054467

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 76 centers in 14 countries.
Groups:
- Pembrolizumab + Epacadostat: Pembrolizumab administered intravenously every 3 weeks. Epacadostat administered orally twice daily.
- EXTREME: EXTREME regimen includes cetuximab + cisplatin or carboplatin + 5-fluorouracil.
  Cetuximab administered intravenously on Cycle 1 Day 1 followed by administration every week. Cisplatin administered intravenously every 3 weeks for </= 6 cycles. Carboplatin administered intravenously every 3 weeks for </= 6 cycles. 5-Fluorouracil administered intravenously every 3 weeks for </= 6 cycles.
Period: Overall Study
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab | EXTREME
Started | 35 | 19 | 35
Intention-to-Treat (ITT) | 35 | 19 | 35
All Participants as Treated (APaT) | 34 | 19 | 34
Completed | 20 | 9 | 19
Not Completed | 15 | 10 | 16
Not completed — Death | 6 | 3 | 10
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — On-going at clinical cut off date | 9 | 6 | 5

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) population consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab | EXTREME | Total
Number analyzed (Participants) | 35 | 19 | 35 | 89
Age, Customized [Mean (Standard Deviation); unit: years] | 62.1 (9.0) | 63.0 (9.6) | 62.7 (10.0) | 62.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 6 | 14
  Male | 30 | 16 | 29 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 34 | 17 | 35 | 86
  Unknown or Not Reported | 1 | 2 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 5 | 13 | 24
  Black Or African American | 1 | 0 | 0 | 1
  White | 28 | 14 | 22 | 64
Primary Tumor Site [Count of Participants; unit: Participants]
  Oropharynx | 12 | 6 | 12 | 30
  Oral Cavity | 10 | 5 | 7 | 22
  Larynx | 9 | 5 | 7 | 21
  Hypopharynx | 4 | 3 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) of Pembrolizumab + Epacadostat, Pembrolizumab Monotherapy and the EXTREME Regimen
Description: ORR was defined as the percentage of participants who had a complete response (CR), disappearance of all target lesions or partial response (PR), >=30% decrease in the sum of the longest diameter of target lesions per RECIST v1.1 by investigator determination.
  Responses are based on investigator assessments per RECIST 1.1 without confirmation using all available scans.
Time Frame: Minimum Week 9
Population: The Intention-to-Treat (ITT) population consisted of all randomized participants.
  The ORR was based on all available imaging assessments after the last participant completed the Week 9 imaging assessment by investigator determination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab | EXTREME
Number analyzed (Participants) | 35 | 19 | 35
percentage of participants | 31.4 [16.9 to 49.3] | 21.1 [6.1 to 45.6] | 34.3 [19.1 to 52.2]

2. Secondary Outcome: Safety and Tolerability of Pembrolizumab + Epacadostat Versus Pembrolizumab Versus the EXTREME Regimen as Measured by Number of Participants Experiencing Adverse Events (AEs)
Description: AE is defined as any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
  Data reported from start of study to data cutoff 17 Jan 2019, up to 14 months.
Time Frame: Up to 14 months
Population: All Participants as Treated (APaT) population consisted of all randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab | EXTREME
Number analyzed (Participants) | 34 | 19 | 34
Participants | 34 | 17 | 34

3. Secondary Outcome: Safety and Tolerability of Pembrolizumab + Epacadostat Versus Pembrolizumab Versus the EXTREME Regimen as Measured by Number of Participants Discontinuing Study Treatment Due to AEs
Description: as for outcome 2
Time Frame: Up to 14 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab | EXTREME
Number analyzed (Participants) | 34 | 19 | 34
Participants | 3 | 2 | 7

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were reported from start of study, up to 30 days after last dose and serious adverse events up to 90 days after last dose are included, up to 14 months
Description: The All Participants as Treated (APaT) population was used for the safety analysis and consisted of all randomized participants who received at least 1 dose of study treatment.
  All-Cause Mortality was based on the ITT population and consisted of all randomized participants.
  MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to the drug are excluded
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab | EXTREME
All-Cause Mortality (participants affected / at risk) | 6/35 | 4/19 | 10/35
Serious Adverse Events (participants affected / at risk) | 12/34 | 8/19 | 12/34
Other Adverse Events (participants affected / at risk) | 34/34 | 17/19 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Epacadostat (N=34) | Pembrolizumab (N=19) | EXTREME (N=34)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Clostridial sepsis (Infections and infestations) | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Epacadostat (N=34) | Pembrolizumab (N=19) | EXTREME (N=34)
Anaemia (Blood and lymphatic system disorders) | 5 | 4 | 19
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 9
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 1 | 0
Hypothyroidism (Endocrine disorders) | 6 | 4 | 1
Eyelid oedema (Eye disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 1
Ankyloglossia acquired (Gastrointestinal disorders) | 0 | 1 | 0
Cheilosis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 1 | 12
Diarrhoea (Gastrointestinal disorders) | 7 | 2 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 2 | 17
Odynophagia (Gastrointestinal disorders) | 2 | 0 | 0
Oral pain (Gastrointestinal disorders) | 2 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 8
Vomiting (Gastrointestinal disorders) | 7 | 0 | 5
Asthenia (General disorders) | 6 | 2 | 8
Chest pain (General disorders) | 2 | 2 | 2
Face oedema (General disorders) | 2 | 1 | 0
Fatigue (General disorders) | 11 | 3 | 7
Malaise (General disorders) | 0 | 0 | 3
Mucosal inflammation (General disorders) | 0 | 0 | 10
Oedema peripheral (General disorders) | 1 | 1 | 1
Pyrexia (General disorders) | 3 | 0 | 5
Swelling (General disorders) | 1 | 1 | 1
Ulcer (General disorders) | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 3
Device related infection (Infections and infestations) | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3 | 3
Oral candidiasis (Infections and infestations) | 1 | 0 | 3
Paronychia (Infections and infestations) | 0 | 0 | 9
Pneumonia (Infections and infestations) | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 5
Amylase increased (Investigations) | 4 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 3 | 1 | 3
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 2
Blood sodium decreased (Investigations) | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1
Lipase increased (Investigations) | 6 | 0 | 4
Lymphocyte count decreased (Investigations) | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 8
Platelet count decreased (Investigations) | 0 | 0 | 12
Weight decreased (Investigations) | 3 | 2 | 8
White blood cell count decreased (Investigations) | 0 | 0 | 7
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 9
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Aphonia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 4
Headache (Nervous system disorders) | 3 | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 5 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 2 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Tracheal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 14
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 0 | 6
Rash (Skin and subcutaneous tissue disorders) | 9 | 4 | 13
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 2 | 3
Hypotension (Vascular disorders) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT03358472/Prot_SAP_000.pdf